CLINICAL TRIAL: NCT05307848
Title: Reproductive Function in Women With Bipolar Disorder: a Prospective Observational Cohort Study
Brief Title: Reproductive Function in Women With Bipolar Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Other Study IDs: RF20220301
Record Dates: First submitted 2022-03-14; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; reproductive function; hormone; menstruation; cognition
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Female patients with bipolar disorder without medication
  Interventions: Other: No intervention
- Female patients with bipolar disorder after stable prescription for ≥6 months
  Interventions: Other: No intervention
- Age and BMI-matched healthy controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Many studies have shown that patients with bipolar disorder are prone to reproductive dysfunction, including polycystic ovary syndrome, hyperprolactinemia, and amenorrhea. However, there is still considerable disagreement about the causes of reproductive dysfunction in patients with bipolar disorder. This study will evaluate the reproductive function of female patients with bipolar disorder without medication and those with bipolar disorder after stable medication, compared with the health control. The purpose of the study is to explore the influence, degree, and possible risk factors of bipolar disorder itself and drugs on the reproductive function of female patients.

DETAILED DESCRIPTION:
This study will comprise 60 female patients with bipolar disorder without medication, 60 female patients with bipolar disorder after stable prescription for ≥6 months, and 60 age and BMI-matched healthy controls. All of whom gave informed consent. All participants will be assessed and clinically examined at baseline, and all patients are encouraged to follow up in the sixth month. Baseline assessments will include demographics, menstrual records, comprehensive medical history, anthropometric measurements (weight and height), physical examination, pelvic ultrasound, and laboratory work (e.g., reproductive hormones). The follow-up of patients will include menstrual records, pelvic ultrasound, and reproductive hormones. Clinical symptoms will be assessed by Hamilton Depression Scale, Hamilton Anxiety Scale, and Young Mania Rating Scale at baseline and week 24. The cognitive function will be assessed at baseline and the sixth month with the Reusable Assessment of Neuropsychological Status Battery (RBANS) and the Stroop Color-Word Test. The primary outcomes will be menstruation, reproductive hormone levels, and pelvic ultrasound. Secondary outcomes will include overall psychiatric symptomatology, quality of life, cognitive function, and other biological data.

ELIGIBILITY:
Inclusion Criteria:

* Test groups：

  1. Subjects voluntarily participated in the trial and signed informed consent and were able to comply with planned visits, laboratory tests, and other study procedures；
  2. Meets the diagnostic criteria for bipolar disorder in the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) and has no coexisting psychiatric disorders；
  3. First diagnosis of bipolar disorder or stable medication for ≥6 months.
* Control group：

  1. Subjects voluntarily participated in the trial and signed informed consent and were able to comply with planned visits, laboratory tests, and other study procedures；
  2. No history of mental illness;
  3. No history of psychotropic medication.

Exclusion Criteria:

1. Presence of any other medical disorder affecting reproductive endocrine function;
2. Taking contraceptives, immunosuppressants, and other drugs that may affect reproductive function within six months;
3. Currently pregnant, breastfeeding, or planning to become pregnant in perimenopause or postmenopause;
4. Those with obvious suicidal tendencies;
5. Serious neurological disease with a clear family history or underlying risk;
6. Combining other severe acute or chronic diseases, mental diseases, or abnormal laboratory tests has clinical significance, and the subject is judged by the investigator to be unsuitable to participate in this study.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Female patients with bipolar disorder without medication, female patients with bipolar disorder after stable prescription for ≥6 months, and BMI-matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in menstrual cycle at baseline and the sixth month | Baseline and the sixth month
Changes in reproductive hormone at baseline and the sixth month | Baseline and the sixth month
Changes in pelvic ultrasonography findings at baseline and the sixth month | Baseline and the sixth month

SECONDARY OUTCOMES:
Change of Hamilton Depression Scale (HAMD) from baseline to the sixth month | Baseline and the sixth month
  Scores ranging from 0-75, with higher scores indicating more severe symptoms
Change of Hamilton Anxiety Scale (HAMA) from baseline to the sixth month | Baseline and the sixth month
  Scores ranging from 0-56, with higher scores indicating more severe symptoms
Change of Young's Mania Scale (YMRS) from baseline to the sixth month | Baseline and the sixth month
  Scores ranging from 0-60, with higher scores indicating more severe symptoms
Change of Reusable Neuropsychological Status Assessment Battery (RBANS) from baseline to the sixth month | Baseline and the sixth month
  Scores ranging from 0-321, with higher scores indicating better cognitive ability

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute of 2nd Xiangya Hospital,CSU, Changsha, China